CLINICAL TRIAL: NCT02426060
Title: Effect of Imrecoxib on the Pharmacokinetics and Pharmacodynamics of Warfarin in Healthy Subjects
Brief Title: A Drug Drug Interaciton Study of Imrecoxib and Warfarin in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARXBDDI-1
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Imrecoxib; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imrecoxib&Warfarin (Experimental)
  Interventions: Drug: Imrecoxib; Drug: Warfarin

INTERVENTIONS:
Drug: Imrecoxib
Drug: Warfarin

SUMMARY:
The objective of this study was to determine the effects of Imrecoxib, an anti-infiammatory/analgesic agent that primarily inhibits COX-2 and not COX-1 at therapeutic doses, on the steady-state pharmacokinetic profile and hypoprothrombinemic effect of warfarin in healthy volunteers.

DETAILED DESCRIPTION:
This is a single center open label study to assess the effect of Imrecoxib on the PK of Warfarin in Healthy Volunteers. The goals of this study are as follows: assess the PK of warfarin when administered alone ,and with Imrecoxib ; assess INR of warfarin when administered alone, and with Imrecoxib; to assess the effect of Imrecoxib on the PK/PD of warfarin, to assess the safety and tolerability of warfarin administered with Imrecoxib.

ELIGIBILITY:
Inclusion Criteria:

Adult males aged 18 to 40 years,with BMI 19~24.

Subjects who, in the opinion of the investigator, are healthy as determined by medical history, physical examination, and 12 Lead ECG.

Willing and able to provide written informed consent.

Exclusion Criteria:

History of hypersensitivity to Imrecoxib and its components.

History or current clinically important systemic illnesses, including but not limited to cardiovascular, pulmonary, hepatobiliary, renal, hematological, gastrointestinal, endocrinological, immunological, dermatological, neurological, or psychiatric diseases, or any conditions that may place the subject at increased risk as determined by the investigator.

Any condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.

History of alcohol dependent, habitual heavy users of caffeinated beverages judged by the investigator.

Have had significant blood loss (>200mL) or have donated 1 or more units of blood or plasma within 12 weeks prior to study entry.

Have a positive test at Screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (HCVAb).

Have used any drugs or substances (including herbal supplements) known to inhibit or induce cytochrome (CYP) P450enzymesincluding CYP3A4, CYP2C8 and CYP2C9 within 4 weeks prior to the first dose and throughout the study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics parameters like Cmax、tmax and AUC0-t of Warfarin | Predose up to 144 hours post Day 1 and Day 10 dose

SECONDARY OUTCOMES:
Prothrombintime after Warfarin dosing | 6 hours to 144 hours post Day 1 and Day10 dose

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital Tongji Medical College Huazhong University of Science and technology, Wuhan, Hubei, China